CLINICAL TRIAL: NCT02032641
Title: Evaluation of Non-Ablative Laser for Treatment of Direct Brow Lift Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sara T. Wester, Ophthalmologist, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20120936
Record Dates: First submitted 2013-06-24; First posted 2014-01-10 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Scar
Keywords: Non-ablative laser; Scar revision; direct brow lift
MeSH Terms: conditions — Cicatrix | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Treatment Side (Experimental): Each patient was randomized to have one of two scars treated with Laser Genesis. The treatment was administered by manually scanning the rapidly pulsed laser in an even, painting motion throughout the entire treatment zone. The eyebrow hairs were covered with white tape to prevent inadvertent alopecia. The laser handpiece was oriented perpendicular to the skin at all times, at a distance of 1-2 cm. Patients were instructed throughout to give verbal feedback regarding if the area was "too hot" as an additional safeguard against epidermal damage.
  Interventions: Device: Laser treatment
- Control side (No Intervention): Each patient had a scar which was randomized to not undergo treatments with Laser Genesis, and was used as a control. Patients were not allowed to undergo laser or any other scar treatments with the exception of sun protection for the control scar for the duration of the study.

INTERVENTIONS:
Device: Laser treatment — Non-ablative, non-fractional, microsecond-pulsed Nd:YAG laser 500-1000 pulses, 0.3 msec pulse duration, 10-14 J/cm2, 5 mm spot size
  Other Names: Laser Genesis, Cutera; 1064 microsecond-pulsed Nd:YAG laser
  Arms: Laser Treatment Side

SUMMARY:
The purpose of this study is to determine the efficacy of the 1064nm Neodymium yttrium aluminum garnet (Nd:YAG) laser (Laser Genesis, Cutera TM) in the treatment of surgical scar after direct brow lift.

DETAILED DESCRIPTION:
Patients who undergo a direct brow lift may participate in this study. Participants will receive laser treatment on one of the two surgical wounds (side of treatment will be chosen randomly by an independent source). Treatment parameters will be 500 spots and 10-14 megajoules (mJ) depending on skin type. The opposite side brow scar will not be treated until 1 month after the study is completed (if the patient elects to treat the contralateral brow after study completion this will be done at no charge to the patient). This treatment will be given at 2-4 week intervals for 6 treatments. Photographs will be taken at each visit, and they will be assessed based on different parameters by an examiner, as well as judged by the patient based on overall appearance.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing or have undergone direct brow lift

Exclusion Criteria:

* under 18 years old
* history of photodermatoses
* receiving systemic isotretinoin within the preceding 6 months
* undergoing other scar treatment in the brow area
* pregnant patients
* history of adverse outcomes related to non-ablative laser

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wester, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Bascom Palmer Eye Institute, Miami, Florida
  - Bascom Palmer Eye Institute, Plantation, Florida

IPD SHARING:
Plan to Share IPD: No
Submitted for publication but no individual participant data released

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients who had undergone direct brow lift within the last three years were contacted by telephone, and an approved script was used for recruitment.
Pre-assignment Details: Exclusion criteria included unilateral procedures, age less than 18 years, pregnancy, history of photodermatoses or adverse outcomes associated with laser, history of isotretinoin use within the prior six months, and active use of other scar treatment in the brow area.
Groups:
- Laser Treatment and Control Group: Each patient was randomized to have one of two scars treated with Laser Genesis and a scar not treated with Laser Genesis, which was used as a control. Patients were not allowed to undergo laser or any other scar treatments with the exception of sun protection for the control scar for the duration of the study. The laser treatment was administered by manually scanning the rapidly pulsed laser in an even, painting motion throughout the entire treatment zone. The eyebrow hairs were covered with white tape to prevent inadvertent alopecia. The laser handpiece was oriented perpendicular to the skin at all times, at a distance of 1-2 cm. Patients were instructed throughout to give verbal feedback regarding if the area was "too hot" as an additional safeguard against epidermal damage.
  Laser treatment: Non-ablative, non-fractional, microsecond-pulsed Neodymium:Yttrium/Aluminum/Garnet laser 500-1000 pulses, 0.3 msec pulse duration, 10-14 J/cm2, 5 mm spot size
Period: Overall Study
Arm/Group | Laser Treatment and Control Group
Started | 9 (18 Brows enrolled for evaluation)
Completed | 8 (16 brows completed study (half underwent treatment, half were control))
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to brows, not participants, as each participant underwent treatment of one brow and the other brow was a control.
Arm/Group | Laser Treatment and Control Group
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Relative Improvement
Description: Which scar, overall, appears to have improved more from initial to final visit, as rated by blinded examiner of photographs
Time Frame: 1 month after final treatment
Population: 3 graders masked to treatments were asked to judge side-by-side photographs of first and final visits for which scar improved more. Each pair of before-and-after photos was graded twice by each examiner. Results are percentage of times treated scar was chosen by examiners as most improved (an analysis of 6 results per pair of photos).
Measure: Mean (Standard Deviation); unit: percentage of times treated scar chosen
Units Other Than Participants: BROW
Groups:
- Control Scar: Each patient had a scar which was randomized to not undergo treatments with Laser Genesis, and was used as a control. Patients were not allowed to undergo laser or any other scar treatments with the exception of sun protection for the control scar for the duration of the study.
Arm/Group | Laser Treatment Side | Control Scar
Number analyzed (Participants) | 8 | 8
Number analyzed (BROW) | 8 | 8
percentage of times treated scar chosen | 50.0 (12.5) | 50.0 (12.5)

2. Secondary Outcome: Overall Appearance
Description: Subjects were asked to rate overall cosmesis of both the treated and control scars on a 1-10 scale, with 1 being extremely poor and 10 being extremely excellent, as rated by participant
Time Frame: 10 minutes before first treatment and at the final visit
Population: Patients were asked to grade overall cosmesis of both the treated and control scars on a 1-10 scale, with 1 being extremely poor and 10 being extremely excellent. Grading was done 10 minutes prior to each laser treatment and 4 weeks after final treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: BROW
Arm/Group | Laser Treatment Side | Control Scar
Number analyzed (Participants) | 8 | 8
Number analyzed (BROW) | 8 | 8
units on a scale
  Before first treatment | 3.75 (2.12) | 4.37 (1.50)
  Final visit | 6.25 (1.98) | 4.50 (2.62)
Statistical Analysis 1: Comparison: Laser Treatment Side; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — The threshold for significance is p<0.05
Statistical Analysis 2: Comparison: Control Scar; Test type: Superiority or Other; p > 0.10, t-test, 1 sided — The threshold for significance is p<0.05

3. Secondary Outcome: Hair Loss
Description: After each laser session, subjects were asked to rate perceived amount of hair loss from both the treated and control scars on a 1-10 scale, with 1 being none at all and 10 being extremely significant
Time Frame: within 1 hour after final treatment
Population: Within 1 hour after treatment, subjects were given a mirror and asked to rate perceived hair loss for each side on a 1-10 scale, with 1 representing none and 10 representing very significant
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: BROW
Arm/Group | Laser Treatment Side | Control Scar
Number analyzed (Participants) | 8 | 8
Number analyzed (BROW) | 8 | 8
units on a scale | 1 (0) | 1 (0)

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Groups:
- Laser Right, Non-laser Left; Laser Left, Non-laser RIght: Group which had the right post-operative scar assigned to receive laser treatment
Arm/Group | Laser Right, Non-laser Left | Laser Left, Non-laser RIght
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No